CLINICAL TRIAL: NCT03837197
Title: Expanded Criteria Donors in Liver and Kidney Transplantation: Protocol of a Randomised Single Center Clinical Trial of Hypothermic Oxygenated Perfusion Versus Static Cold Storage
Brief Title: Clinical Trial of New Hypothermic Oxygenated Perfusion System Versus Static Cold Storage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Matteo Ravaioli, MD, Principal Investigator, General Manager of General Surgery, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RF-2016-02364732
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Liver Diseases; Kidney Diseases
Keywords: donors and donation; Extended criteria donor; Organ perfusion and preservation; Liver transplantation; Kidney transplantation; Preservation injury; Ischemia reperfusion injury
MeSH Terms: conditions — Liver Diseases; Kidney Diseases; Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kidney-Hypothermic oxygenated (Experimental): Belzer machine perfusion solution at 4°C-10°C in sterile conditions and continuous oxygenation (partial pressure of oxygen=500-600 mmHg) will be used for perfusion 2000 ml for kidneys.
  Interventions: Device: Kidney-Hypothermic oxygenated
- Kidney-Static Cold Storage (No Intervention): Kidneys undergoing SCS will be stored in sterile organ bags with Celsior or University of Wisconsin solution and cooled in ice.
- Liver-Hypothermic oxygenated (Experimental): Belzer machine perfusion solution at 4°C-10°C in sterile conditions and continuous oxygenation (partial pressure of oxygen=500-600 mmHg) will be used for perfusion 3000 ml for livers.
  Interventions: Device: Liver-Hypothermic oxygenated
- Liver-Static Cold Storage (No Intervention): Livers undergoing SCS will be stored in sterile organ bags with Celsior or University of Wisconsin solution and cooled in ice.

INTERVENTIONS:
Device: Kidney-Hypothermic oxygenated — Kidney perfusion will be performed through the renal artery at 25-30 mmHg pressure.
  Flow, pressure and temperature will be monitored and registered on a Universal Serial Bus (USB) memory system during organ perfusion. Gas analysis of the effluent perfusate will be accomplished at the start of perfusion (T0) then every 30 minutes. Two perfusate samples will be collected at the beginning and at the end of perfusion to rule out bacterial or fungal contamination.
  HOPE will start by flushing the organ at low flow values (20 ml/min) with new oxygenated perfusion fluid during back-table preparation. Organ will be treated with continuous HOPE until transplant. Organ perfusion will be continuously monitored. Minimal perfusion time will be 2 hours for kidneys.
  Arms: Kidney-Hypothermic oxygenated
Device: Liver-Hypothermic oxygenated — Liver perfusion will be performed through the portal vein at a 5 mmHg pressure.
  Flow, pressure and temperature will be monitored and registered on a Universal Serial Bus (USB) memory system during organ perfusion. Gas analysis of the effluent perfusate will be accomplished at the start of perfusion (T0) then every 30 minutes. Two perfusate samples will be collected at the beginning and at the end of perfusion to rule out bacterial or fungal contamination.
  HOPE will start by flushing the organ at low flow values (30 ml/min) with new oxygenated perfusion fluid during back-table preparation. Organ will be treated with continuous HOPE until transplant. Organ perfusion will be continuously monitored. Minimal perfusion time will be 1 hour for livers.
  Arms: Liver-Hypothermic oxygenated

SUMMARY:
With the present study the investigators will evaluate the benefit of end-ischemic HOPE on ECD grafts (livers and kidneys) as compared to SCS. Organs will be perfused through a recently developed machine perfusion (MP) device, from the beginning of back-table procedures till implantation, without increasing CIT. The aim of the study will be demonstrating the ability of HOPE to improve graft function and post-operative outcomes of ECD kidney and liver recipients.

DETAILED DESCRIPTION:
Extended criteria donors (ECD) are widely utilized due to organ shortage, but this may increase the risk of graft dysfunction and of poorer outcomes.

Hypothermic oxygenated perfusion (HOPE) is a recent organ preservation strategy for marginal kidney and liver grafts, which allows to redirect anaerobic metabolism to aerobic metabolism under hypothermic conditions and to protect grafts from oxidative species-related damage; these mechanisms may potentially improve graft function and survival.

Methods This is an open-label, randomized multicenter clinical trial with the aim of comparing HOPE vs. static cold storage (SCS) in ECD kidney and liver transplantation.

In the study protocol - approved by ethics committee - 220 patients (110 liver recipients and 110 kidney recipients) will be enrolled. Livers and kidneys assigned to HOPE will be perfused by machine perfusion with cold Belzer solution (4°-10°C) and with continuous oxygenation (partial pressure of oxygen = 500-600 mmHg). In the control group, livers and kidneys undergoing SCS will be steeped in Celsior or University of Wisconsin Belzer solutions and stored in ice. Using the same perfusion machine for both liver and kidney grafts, organs will be perfused from the start of the back-table procedure until implantation, without increasing cold ischemia time (CIT). For each group the investigators will evaluate clinical outcomes, graft function tests and histologic findings, as well as perfusate and the number of allocated organs.

ELIGIBILITY:
Inclusion Criteria:

* For kidneys: donor age ≥ 60 years or 50-59 years with two or more of the sequent risk factors: death due to cerebrovascular accident, history of hypertension, donor serum creatinine > 1.5 mg/dL, cold ischemia time (CIT) > 20 h;
* For livers: donors with hemodynamic deterioration, donor age > 65 years, donor body mass index > 30 kg/m2, serum bilirubin > 3 mg/dl, AST or ALT above three times the upper reference threshold, sodium > 165 mmol/l, intensive care unit (ICU) stay > 7 days, steatosis > 40%, CIT > 12 h.

Exclusion Criteria:

* Donor age ≤18 years;
* Donors after circulatory death (DCD) will be excluded, because Italian law requires 20 minutes of "no touch period" before death declaration, causing prolonged warm ischemia and subsequent mandatory perfusion of the organ.
* Split-liver recipients, liver transplantation (LT) for acute liver failure, pre-emptive renal transplant, dual kidney transplantation, and patients with intra-operative surgical complications before the organ implantation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Liver Transplant - Early allograft dysfunction (EAD) | 0-30 days after procedure
  Present/Non present
Kidney Transplant- Delayed graft function (DGF) | 0-30 days after procedure
  Present/Non present

SECONDARY OUTCOMES:
Liver and Kidney surgical complications | 0-6 months after procedure
  Present/Non present
Liver and Kidney graft function at 6 and 12 months | 0-12 months after procedure
  Functioning/non functioning
Patient survival at 6 and 12 months | 0-12 months after procedure
  Alive/Death

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Ravaioli, PhD, Principal Investigator — University of Bologna S.Orsola-Malpighi Hospital
Locations (1):
- Azienda Ospedaliera di Bologna - Policlinico S. Orsola Malpighi, Bologna, Italy

REFERENCES:
- [Background] Belzer FO, Southard JH. Principles of solid-organ preservation by cold storage. Transplantation. 1988 Apr;45(4):673-6. doi: 10.1097/00007890-198804000-00001. No abstract available. PMID 3282347
- [Background] Tanrisev M, Hoscoskun C, Asci G, Sozbilen M, Firat O, Ertilav M, Ozkahya M, Toz H. Long-term outcome of kidney transplantation from elderly living and expanded criteria deceased donors. Ren Fail. 2015 Mar;37(2):249-53. doi: 10.3109/0886022X.2014.982488. Epub 2014 Dec 3. PMID 25470081
- [Background] Feng S, Goodrich NP, Bragg-Gresham JL, Dykstra DM, Punch JD, DebRoy MA, Greenstein SM, Merion RM. Characteristics associated with liver graft failure: the concept of a donor risk index. Am J Transplant. 2006 Apr;6(4):783-90. doi: 10.1111/j.1600-6143.2006.01242.x. PMID 16539636
- [Background] Ravaioli M, Baldassare M, Vasuri F, Pasquinelli G, Laggetta M, Valente S, De Pace V, Neri F, Siniscalchi A, Zanfi C, Bertuzzo VR, Caraceni P, Trere D, Longobardi P, Pinna AD. Strategies to Restore Adenosine Triphosphate (ATP) Level After More than 20 Hours of Cold Ischemia Time in Human Marginal Kidney Grafts. Ann Transplant. 2018 Jan 12;23:34-44. doi: 10.12659/aot.905406. PMID 29326416
- [Background] Ravaioli M, De Pace V, Comai G, Busutti M, Del Gaudio M, Amaduzzi A, Cucchetti A, Siniscalchi A, La Manna G, D'Errico AAD, Pinna AD. Successful Dual Kidney Transplantation After Hypothermic Oxygenated Perfusion of Discarded Human Kidneys. Am J Case Rep. 2017 Sep 20;18:1009-1013. doi: 10.12659/ajcr.905377. PMID 28928357
- [Background] Kron P, Schlegel A, de Rougemont O, Oberkofler CE, Clavien PA, Dutkowski P. Short, Cool, and Well Oxygenated - HOPE for Kidney Transplantation in a Rodent Model. Ann Surg. 2016 Nov;264(5):815-822. doi: 10.1097/SLA.0000000000001766. PMID 27584571
- [Background] Schlegel A, Muller X, Dutkowski P. Hypothermic Machine Preservation of the Liver: State of the Art. Curr Transplant Rep. 2018;5(1):93-102. doi: 10.1007/s40472-018-0183-z. Epub 2018 Jan 22. PMID 29564206
- [Background] Dutkowski P, Polak WG, Muiesan P, Schlegel A, Verhoeven CJ, Scalera I, DeOliveira ML, Kron P, Clavien PA. First Comparison of Hypothermic Oxygenated PErfusion Versus Static Cold Storage of Human Donation After Cardiac Death Liver Transplants: An International-matched Case Analysis. Ann Surg. 2015 Nov;262(5):764-70; discussion 770-1. doi: 10.1097/SLA.0000000000001473. PMID 26583664
- [Background] Port FK, Bragg-Gresham JL, Metzger RA, Dykstra DM, Gillespie BW, Young EW, Delmonico FL, Wynn JJ, Merion RM, Wolfe RA, Held PJ. Donor characteristics associated with reduced graft survival: an approach to expanding the pool of kidney donors. Transplantation. 2002 Nov 15;74(9):1281-6. doi: 10.1097/00007890-200211150-00014. PMID 12451266
- [Background] Attia M, Silva MA, Mirza DF. The marginal liver donor--an update. Transpl Int. 2008 Aug;21(8):713-24. doi: 10.1111/j.1432-2277.2008.00696.x. Epub 2008 May 19. PMID 18492121
- [Background] Ravaioli M, De Pace V, Comai G, Capelli I, Baraldi O, D'Errico A, Bertuzzo VR, Del Gaudio M, Zanfi C, D'Arcangelo GL, Cuna V, Siniscalchi A, Sangiorgi G, La Manna G. Preliminary experience of sequential use of normothermic and hypothermic oxygenated perfusion for donation after circulatory death kidney with warm ischemia time over the conventional criteria - a retrospective and observational study. Transpl Int. 2018 Nov;31(11):1233-1244. doi: 10.1111/tri.13311. Epub 2018 Jul 20. PMID 29957863
- [Background] Olthoff KM, Kulik L, Samstein B, Kaminski M, Abecassis M, Emond J, Shaked A, Christie JD. Validation of a current definition of early allograft dysfunction in liver transplant recipients and analysis of risk factors. Liver Transpl. 2010 Aug;16(8):943-9. doi: 10.1002/lt.22091. PMID 20677285
- [Background] Agopian VG, Harlander-Locke MP, Markovic D, Dumronggittigule W, Xia V, Kaldas FM, Zarrinpar A, Yersiz H, Farmer DG, Hiatt JR, Busuttil RW. Evaluation of Early Allograft Function Using the Liver Graft Assessment Following Transplantation Risk Score Model. JAMA Surg. 2018 May 1;153(5):436-444. doi: 10.1001/jamasurg.2017.5040. PMID 29261831
- [Background] Humar A, Ramcharan T, Kandaswamy R, Gillingham K, Payne WD, Matas AJ. Risk factors for slow graft function after kidney transplants: a multivariate analysis. Clin Transplant. 2002 Dec;16(6):425-9. doi: 10.1034/j.1399-0012.2002.02055.x. PMID 12437622
- [Background] Schlegel A, de Rougemont O, Graf R, Clavien PA, Dutkowski P. Protective mechanisms of end-ischemic cold machine perfusion in DCD liver grafts. J Hepatol. 2013 Feb;58(2):278-86. doi: 10.1016/j.jhep.2012.10.004. Epub 2012 Oct 11. PMID 23063573
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597
- [Result] Versteilen AM, Di Maggio F, Leemreis JR, Groeneveld AB, Musters RJ, Sipkema P. Molecular mechanisms of acute renal failure following ischemia/reperfusion. Int J Artif Organs. 2004 Dec;27(12):1019-29. doi: 10.1177/039139880402701203. PMID 15645611
- [Derived] Ravaioli M, Germinario G, Dajti G, Sessa M, Vasuri F, Siniscalchi A, Morelli MC, Serenari M, Del Gaudio M, Zanfi C, Odaldi F, Bertuzzo VR, Maroni L, Laurenzi A, Cescon M. Hypothermic oxygenated perfusion in extended criteria donor liver transplantation-A randomized clinical trial. Am J Transplant. 2022 Oct;22(10):2401-2408. doi: 10.1111/ajt.17115. Epub 2022 Jun 21. PMID 35671067
- [Derived] Ravaioli M, Maroni L, Angeletti A, Fallani G, De Pace V, Germinario G, Odaldi F, Corradetti V, Caraceni P, Baldassarre M, Vasuri F, D'Errico A, Sangiorgi G, Siniscalchi A, Morelli MC, Rossetto A, Ranieri VM, Cescon M, Del Gaudio M, Zanfi C, Bertuzzo V, Comai G, La Manna G. Hypothermic Oxygenated Perfusion Versus Static Cold Storage for Expanded Criteria Donors in Liver and Kidney Transplantation: Protocol for a Single-Center Randomized Controlled Trial. JMIR Res Protoc. 2020 Mar 19;9(3):e13922. doi: 10.2196/13922. PMID 32191209
- See also: Sistema Informativo Trapianti (SIT) — https://trapianti.sanita.it